CLINICAL TRIAL: NCT01813851
Title: Effect of Intradialytic Physical ACTIvity in Addition to a NUTritional Support on Protein Energy Wasting and Physical Functioning in Chronic Hemodialysis Patients ("ACTINUT" Study), Multicenter, Randomized, Controlled Open Label Trial Study Multicenter, Prospective, Randomized Study
Brief Title: Effect of Intradialytic Physical ACTIvity in Addition to a NUTritional Support on Protein Energy Wasting and Physical Functioning in Chronic Hemodialysis Patients ("ACTINUT" Study)
Acronym: ACTINUT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC12_0487
Record Dates: First submitted 2013-03-12; First posted 2013-03-19 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Renal Failure, Hemodialysis Treatment, Protein-energy Wasting
Keywords: Dialysis, Exercise, Protein Energy Wasting, Nutrition and Physical Fitness
MeSH Terms: conditions — Kidney Failure, Chronic; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (No Intervention): Patients in the "control group" will receive:
  Dietary counseling by a dietician and if necessary modification of the prescription of oral nutritional supplements or intradialytic parenteral nutrition to reach recommended targets according to the European Best Practice Guidelines on Nutrition (energy intake 30-40 kcal/kg of ideal weight/day, protein intake 1.1 g/kg of ideal weight/day
- activity group (Experimental): Patients in the "group exercise" will:
  Dietary counseling by a dietician and if necessary modification of the prescription of oral nutritional supplements or intradialytic parenteral nutrition to reach recommended targets according to the European Best Practice Guidelines on Nutrition (energy intake 30-40 kcal/kg of ideal weight/day, protein intake 1.1 g/kg of ideal weight/day A program of physical activity consisting of progressive endurance and resistance training on a cycle ergometer, performed during the dialysis session under supervision and counseling by a qualified trainer
  Interventions: Device: Exercise training in addition to nutritional support

INTERVENTIONS:
Device: Exercise training in addition to nutritional support
  Other Names: Reck MOTOmed® Letto
  Arms: activity group

SUMMARY:
Sedentary behavior and protein-energy wasting (PEW) are well known risk factors of adverse outcome and low quality of life in chronic renal failure patients treated by dialysis. Treatment strategies of PEW by different types of nutritional support (as dietary counseling, oral nutritional supplements or intradialytic parenteral nutrition) have limited efficacy. Physical activity has been shown to have numerous positive impacts in pathologic conditions associated to end stage renal disease.

Concomitant prescription of physical activity and nutritional support might mutually enhance the anabolic effects of these interventions and improve the rate of remission of PEW.

The aim of this study is to analyze the effect of a programmed, progressive endurance training performed during the dialysis session on a cycle ergometer under the supervision of a qualified trainer, on protein energy wasting and physical functioning of chronic hemodialysis patients.

DETAILED DESCRIPTION:
Aim 1: To determine the percentage of patients in remission from the state of protein- energy wasting. Hypothesis 1: Patients in the exercise group will more frequently reverse the PEW than in the control group Aim 2: To determine the patterns of change in body composition (fat free mass). Hypothesis 2: Patients in the exercise group will maintain or increase their fat free mass and patients in the control group will decrease their fat free mass Aim 3: To determine the effects of exercise on muscle strength. Hypothesis 3: Patients in the exercise group will maintain or increase their quadriceps strength while patients in the control group will decrease their muscle strength Aim 4: To determine the effects of exercise on postural balance. Hypothesis 4: Patients in the exercise group will maintain or increase their body balance while patients in the control group will decrease their body balance Aim 5: To determine the effects of exercise on quality of life as assessed by the SF-36. Hypothesis 5: Patients in exercise group will maintain or increase their quality of life form while patients in the control group will decrease their quality of life

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years, treated by hemodialysis since more than 3 months
* Patients considered to be in a clinical stable state, defined as the absence of acute disease or hospitalization during the last month prior to study begin
* Patients fulfilling the diagnostic criteria of protein energy wasting according to the definition proposed by the International Society of Renal Nutrition and Metabolism (ISRNM)
* Patients having signed the informed consent for the study participation
* Patients covered by medical insurance

Exclusion Criteria:

* Medical contraindication or inability to perform physical exercise
* Inadequate dialysis (KT/V< 1.2)
* Poor hemodynamic tolerance of dialysis
* Systemic inflammation (CRP >20 mg/l)
* Pregnancy
* Major trust

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Number of patients who correct the state of protein energy wasting in intervention group compared to a control group | at 6 months

SECONDARY OUTCOMES:
Body composition (fat free mass), assessed by bioimpedance spectroscopy using the Body composition monitor (BCM) | at 3 months and at 6 months
Quadriceps strength measured by dynamometer | at 3 months and at 6 monts
Performance (distance and velocity) in the 6 minute walk test | at 3 months and 6 months
Postural balance as measured by a force platform | at 3 months and at 6 months
Quality of life as measured by the SF-36 test | at the 3 months and at 6 months
The number of hospitalization days | at the 3 months and the 6 months
The survival | at the 3 months and at the 6 months
The dosage of albumin | at the 3 months and at the 6 months
The dosage of prealbumin | at 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dan Hristea, Dr, Principal Investigator — ECHO
Locations (2):
- France (2):
  - ECHO center ( confluent site ), Nantes
  - ECHO CENTER( St-Jacques), Nantes

REFERENCES:
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639
- [Derived] Mah JY, Choy SW, Roberts MA, Desai AM, Corken M, Gwini SM, McMahon LP. Oral protein-based supplements versus placebo or no treatment for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2020 May 11;5(5):CD012616. doi: 10.1002/14651858.CD012616.pub2. PMID 32390133
- [Derived] Magnard J, Deschamps T, Cornu C, Paris A, Hristea D. Effects of a six-month intradialytic physical ACTIvity program and adequate NUTritional support on protein-energy wasting, physical functioning and quality of life in chronic hemodialysis patients: ACTINUT study protocol for a randomised controlled trial. BMC Nephrol. 2013 Nov 26;14:259. doi: 10.1186/1471-2369-14-259. PMID 24279747